CLINICAL TRIAL: NCT00733239
Title: Drug Discrimination in Methadone-Maintained Humans Study 2
Acronym: OMDD2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: R01DA010017-02 (NIH); R01DA010017-02 (NIH); 104881; 5R01DA010017-02 (NIH); DPMCDA
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Opioid Dependence
Keywords: methadone; opioid dependence; opioid
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Diltiazem; Gabapentin; Isradipine; Nifedipine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Receives 2-4 of the drugs listed under Intervention
  Interventions: Drug: 2-4 of the drugs listed below

INTERVENTIONS:
Drug: 2-4 of the drugs listed below — Cycloserine: 500, 675, 750 mg oral capsule may possibly be given Diltiazem: 30, 60, 120 mg oral capsule may possibly be given Gabapentin: 100, 200, 400 mg oral capsule may possibly be given Isradipine: 5, 10 mg oral capsule may possibly be given Naloxone: 0.15 mg/70 kg or 0.2 mg I.M. injection may possibly be given Nifedipine: 5, 10, 20 mg oral capsule may possibly be given Placebo (sugar pill or microcrystalline cellulose): oral capsule may possibly be given Saline: I.M. injection may possibly be given Verapamil: 30, 60, 120 mg oral capsule may possibly be given
  Other Names: Cycloserine: Calan, Veralan; Diltiazem: Cardizem; Gabapentin: Neurontin; Isradipine: DynaCirc; Naloxone: Narca; Nifedipine: Adalat, Procardia; Placebo; Saline; Verapamil: Veralan

SUMMARY:
This study involves giving psychoactive drugs intramuscularly (injected into the muscle of the upper arm or the hip) and/or orally, and measuring the subject's ability to tell the difference between one drug and another, as well as measuring the effects of the drugs on mood, physiology (e.g., heart rate, blood pressure, respiration rate) and behavior. Each subject will receive 2-4 of the listed interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between the ages of 18-65.
2. Participation in the UAMS Substance Abuse Treatment Clinic Methadone Maintenance Program or the Catar Clinic Little Rock with maintenance on a stable dose of methadone (+ or - 10 mg) for at least 1 month prior to study entry.
3. Subjects would have to be in "good standing" in the methadone maintenance program in order to participate; i.e., compliance with scheduled medication and group therapy session hours. This would be defined as < 3 missed methadone medications and missed < 3 group or <3 individual therapy sessions in the month prior to study participation
4. Subjects must submit a urine sample negative for illicit drugs prior to study entry.
5. Subjects must be able to read and understand English.

Exclusion Criteria:

1. Unstable medical condition or stable medical condition that would interact with study medications or participation.
2. Current diagnosis of other drug or alcohol physical dependence (other than tobacco).
3. History of major psychiatric disorder (psychosis, schizophrenia, bipolar, depression)
4. Pregnancy, plans to become pregnant or inadequate birth control.
5. Present or recent (< 1 week) use of over-the-counter psychoactive drug, prescription psychoactive drug or drug that would have major interaction with drugs to be tested. Recent use will be defined based upon the pharmacokinetics of the drug and dosing schedule. Thus, a short-acting antihistamine taken as needed (e.g., once the night before) will not necessarily rule out a participant; however,
6. History of severe reaction to Narcan challenge, which may have been given as part of admission into the Methadone Maintenance Program or to reverse overdose.
7. Liver function tests (ALT, AST) greater than 3 times normal, BUN and Creatinine outside normal range, or thyroid function tests outside normal range.
8. ECG abnormalities including but not limited to: bradycardia (<60 bpm); Wolff-Parkinson White syndrome; wide complex tachycardia; 2nd degree, Mobitz type II heart block; 3rd degree heart block; left or right bundle branch block.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Drug Discrimination Performance | Every Session

SECONDARY OUTCOMES:
Self-report Ratings | Every Session
Vital Signs | Every Session
ECG | Test Sessions

CONTACTS AND LOCATIONS:
Overall Officials: Alison Oliveto, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Fitzgerald LR, Stanley NC, Guise JB, Cargile CS, Mancino MJ, Oliveto AH. Gabapentin and D-cycloserine alone and in combination with naloxone in methadone-maintained humans responding under a naloxone novel-response discrimination procedure. Behav Pharmacol. 2025 Aug 1;36(5):265-275. doi: 10.1097/FBP.0000000000000823. Epub 2025 Apr 8. PMID 40272204